CLINICAL TRIAL: NCT03802396
Title: Modulating ApoE Signalling to Reduce Brain Inflammation, deLirium and postopErative Cognitive Dysfunction (MARBLE): A Phase 2 Trial to Evaluate the Efficacy and Feasibility of CN-105 in Preventing Postoperative Cognitive Dysfunction and Delirium
Brief Title: Modulating ApoE Signalling to Reduce Brain Inflammation, deLirium and postopErative Cognitive Dysfunction
Acronym: MARBLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Miles Berger, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Miles Berger, MD PhD, Assistant Professor, Neuroanesthesiology Division, Anesthesiology Department, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00088855
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: Delirium; Aging; Elderly; Postoperative; Cognitive Dysfunction
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Delirium; Cognitive Dysfunction | interventions — apolipoprotein E mimetic peptide CN-105

STUDY DESIGN:
Intervention Model Description: Investigators will enroll 201 patients total in this phase 2 escalating dose study, with escalating CN-105 doses occurring in three successive groups of 67 patients each. In each group of 67 patients, 50 will receive a given dose of CN-105 and 17 will receive placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to receive either CN-105 or placebo after they consent to participate in the trial. Participants will be enrolled in 1 of 3 dose cohorts of 67 subjects each. An independent statistician will prepare dose stratified mixed block size randomization lists in a 3 to 1 ratio to achieve the desired distribution of drug and placebo. In each block of 67 trial participants, 50 will receive CN-105 and 17 will receive placebo, in a double-blind fashion.
  CN-105 and placebo will be prepared in identical bags labelled simply with the trial participant's number (1-201) to keep all trial staff and clinicians blinded to randomization. Only the investigational pharmacist will have the randomization list for each participant showing what dose of CN-105 or placebo will be administered. To minimize bias, investigators conducting the laboratory assays on the CSF and blood samples will be blinded to trial group assignment during the course of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CN-105 (Experimental): Cohort 1: 50 Patients Dose of CN-105: 0.1 mg/kg
  Cohort 2: 50 Patients Dose of CN-105: 0.5 mg/kg
  Cohort 3: 50 Patients Dose of CN-105: 1 mg/kg
  Interventions: Drug: CN-105
- Placebo (Placebo Comparator): Cohort 1: 17 Patients receiving placebo
  Cohort 2: 17 Patients receiving placebo
  Cohort 3: 17 Patients receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CN-105 — Three doses of CN-105 will be used in three successive cohorts of 50 patients each.
  0.1 mg/kg (cohort 1), 0.5 mg/kg (cohort 2), 1 mg/kg (cohort 3)
  The study drug will be administered by IV every 6 hours, beginning 1 hour prior to surgery, until postoperative day 3 or hospital discharge, whichever occurs first, up to a maximum of 13 doses.
  Arms: CN-105
Drug: Placebo — Patients will receive placebo intravenously every 6 hours, beginning 1 hour prior to surgery, until postoperative day 3 or hospital discharge, whichever occurs first, up to a maximum of 13 doses, identical to those receiving the study drug.
  Arms: Placebo

SUMMARY:
This research study will evaluate the effectiveness and estimate the feasibility of administering an investigational drug called 'CN-105' (the study drug), to prevent postoperative cognitive decline, delirium (serious confusion) and underlying brain inflammatory and brain activity changes in adults 60 years and older undergoing surgery.

DETAILED DESCRIPTION:
This research study will evaluate the effectiveness and estimate the feasibility of administering an investigational drug called 'CN-105' (the study drug), to prevent postoperative cognitive decline, delirium (serious confusion) and underlying brain inflammatory and brain activity changes in adults 60 years and older undergoing surgery. The word "investigational" means the study drug is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA).

It is hoped that CN-105 will block signaling via a gene known as ApoE4, the most common gene implicated in late life Alzheimer's disease.

Depending on when patients enroll in this study, participants will receive either a placebo or a progressively higher dose of CN-105 until the safest and best tolerated dose is reached. The study drug is given via IV (intravenous, meaning through a vein) infusion in the hospital. Study drug infusions will be given up to 4 days after surgery.

Participants will also perform memory and thinking tests, as well as complete a survey and functional assessments, both prior to surgery and again 6 weeks after surgery. Each of those research visits will last about 1 hour.

Additionally, the investigators will collect a blood sample and a cerebrospinal fluid (CSF) sample prior to the participant's surgery, 24 hours after surgery, and again 6 weeks after surgery. To obtain the CSF (cerebrospinal fluid) sample, investigators will perform a lumbar (the lower part of the spinal column) puncture. During surgery, investigators will also record participant brain waves from the scalp using an EEG (electroencephalography) monitor. An electroencephalography monitor reads the electrical activity of the brain in different places using a cap with sensors that is worn on the head.

Although previous studies have not found any associations between the study drug and any serious medical problems, investigators will monitor its effect on wound healing and postoperative infections.

Benefits of this study include the possibility of fewer problems in thinking and memory after surgery if this study drug works as hoped.

Risks of participation in this study include headache, infection/discomfort from the lumbar puncture, discomfort from the blood draw, and minor skin irritation or redness from the EEG and heart rate monitor procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60
* Ability to speak English
* Undergoing non-cardiac, non-neurologic surgical procedures; surgery scheduled to last > 2 hours; due to be admitted to the hospital following surgery

Exclusion Criteria:

* Inmate of a correctional facility
* Scheduled to receive systemic chemotherapy between the time of the two cognitive testing sessions
* Known inability to undergo LPs due to anticoagulant use, severe anxiety, or other clinical contraindication known ahead of time.
* Inappropriate for study inclusion based on the judgement of the principal investigator.
* If a patient undergoes major head trauma that occurs between the times of the two cognitive testing sessions, then they will be withdrawn from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CN-105: The study drug will be administered by IV every 6 hours, beginning 1 hour prior to surgery, until postoperative day 3 or hospital discharge, whichever occurs first, up to a maximum of 13 doses.
Period: Overall Study
Arm/Group | CN-105 | Placebo
Started | 140 | 49
Completed | 137 | 49
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Surgery Cancelled | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CN-105 | Placebo | Total
Number analyzed (Participants) | 137 | 49 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (5.0) | 69.5 (6.0) | 68.7 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 16 | 67
  Male | 86 | 33 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 135 | 47 | 182
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 122 | 42 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 137 | 49 | 186

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs) of Grade II or Higher Per Patient
Description: Safety of CN-105 administration, as measured by adverse event (AE) rates of Grade II and higher in CN-105 versus placebo-treated patients.
Time Frame: up to 6-week follow-up
Population: Participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: events per participant
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 137 | 49
events per participant | 1 [1 to 3] | 2 [1 to 5]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Test type: Other; p = 0.025, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Cerebrospinal Fluid (CSF) IL-6 Cytokine Levels Between Drug vs Placebo Treated Patients
Description: Change in CSF IL-6 cytokine levels from before to after surgery between drug vs placebo treated patients.
Time Frame: Baseline, 24 hours, approximately 6 weeks
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 137 | 49
pg/mL
  Baseline to 24 hours: number analyzed (Participants) | 98 | 37
  Baseline to 24 hours | 0.52 [-0.08 to 1.35] | 0.91 [0.30 to 1.63]
  Baseline to 6 weeks: number analyzed (Participants) | 51 | 20
  Baseline to 6 weeks | -0.06 [-0.40 to 0.17] | 0.00 [-0.20 to 0.12]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Baseline to 24 hours; Test type: Other; p = 0.116, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CN-105 vs Placebo; Baseline to 6 weeks; Test type: Other; p = 0.388, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in CSF IL-8 Cytokine Levels Between Drug vs Placebo Treated Patients
Description: Change in CSF IL-8 cytokine levels from before to after surgery between drug vs placebo treated patients
Time Frame: Baseline, 24 hours, approximately 6 weeks
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 98 | 37
pg/mL
  Baseline to 24 hours | 130.11 [69.11 to 227.90] | 153.43 [67.44 to 268.26]
  Baseline to 6 weeks: number analyzed (Participants) | 51 | 20
  Baseline to 6 weeks | -2.7 [-8.06 to 0.32] | 0.54 [-4.23 to 4.08]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Baseline to 24 hours; Test type: Other; p = 0.569, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CN-105 vs Placebo; Baseline to 6 weeks; Test type: Other; p = 0.047, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in CSF MCP-1 Cytokine Levels Between Drug vs Placebo Treated Patients
Description: Change in CSF MCP-1 cytokine levels before to after surgery between drug vs placebo treated patients
Time Frame: Baseline, 24 hours, approximately 6 weeks
Population: Participants with data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 98 | 37
pg/mL
  Baseline to 24 hours | -114.39 [-177.58 to -22.06] | -116.75 [-195.11 to -26.95]
  Baseline to 6 weeks: number analyzed (Participants) | 51 | 20
  Baseline to 6 weeks | -17.69 [-58.01 to 21.33] | -4.62 [-32.16 to 6.32]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Baseline to 24 hours; Test type: Other; p = 0.498, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CN-105 vs Placebo; Baseline to 6 weeks; Test type: Other; p = 0.745, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in CSF G-CSF Cytokine Levels Between Drug vs Placebo Treated Patients
Description: Change in CSF G-CSF cytokine levels before to after surgery between drug vs placebo treated patients.
Time Frame: Baseline, 24 hours, approximately 6 weeks
Population: Participants who had data collected at each timepoint.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 98 | 37
pg/mL
  Baseline to 24 hours | 2.46 [0.75 to 6.36] | 3.3 [1.89 to 10.18]
  Baseline to 6 weeks: number analyzed (Participants) | 51 | 20
  Baseline to 6 weeks | 0.22 [-1.10 to 1.13] | -0.23 [-0.96 to 0.77]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Baseline to 24 hours; Test type: Other; p = 0.177, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: CN-105 vs Placebo; Baseline to 6 weeks; Test type: Other; p = 0.478, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Cognitive Change Index (CCI) Between Drug vs Placebo Treated Patients
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a Z-score standardization was performed on the 11 cognitive test scores with mean and standard deviation derived at the baseline timepoint. We then constructed four summary scores by taking the average of the standardized cognitive test scores, which represent the following cognitive domains: verbal memory, executive function, visual memory and attention. To quantify overall cognitive function, a cognitive index was calculated as the mean of the 4 domain scores. The cognitive index score has a mean of zero, thus any positive score is above the mean, any negative score is below the mean. A continuous change score was then calculated by subtracting the baseline from the 6-week cognitive index. The resulting outcome measure is unbounded with standard deviation of 0.33. A negative change score indicating decline and a positive score indicating improvement.
Time Frame: Baseline, approximately 6 weeks
Population: Participants who completed both baseline and 6-week follow-up visit and surgery on protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 108 | 35
units on a scale | 0.08 (0.33) | 0.06 (0.34)
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Test type: Other; p = 0.803, t-test, 2 sided

7. Secondary Outcome: Feasibility of Drug Administration as Measured by the Percentage of Doses Given Within the Correct Time Window
Description: The feasibility of perioperative CN-105 administration is assessed by tracking the percentage of doses given within the correct time window (i.e. within 1 hour prior to the scheduled or actual start time of the surgery, and within a +/- 90 minute time window for subsequent doses, which are administered every 6 hours after the start of surgery).
Time Frame: admission to preoperative holding to hospital discharge (up to postoperative day 4)
Measure: Mean (95% Confidence Interval); unit: percentage of doses
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 137 | 49
percentage of doses | 94.6 [92.9 to 96.0] | 93.8 [90.8 to 96.0]

8. Secondary Outcome: Number of Participants Who Experience Delirium
Description: Scores on 3D CAM (non-intubated patients) or CAM ICU (intubated patients) are used to determine whether patients have delirium (yes/no).
Time Frame: Baseline, day of surgery (twice), post-operative days 1 - 5 (twice), 6 weeks +/- 3 weeks
Population: Participants who completed surgery on protocol and had at least 1 postoperative CAM-3D or CAM-ICU assessment performed.
Measure: Count of Participants; unit: Participants
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 135 | 49
Participants | 26 | 13
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Test type: Other; p = 0.286, Chi-squared; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.41 to 1.30]

9. Secondary Outcome: Peak Severity of Delirium Symptoms Between Drug vs. Placebo Treated Patients
Description: Scores on the 3D CAM (in non-intubated patients) are used to determine delirium symptom severity based on a 0 - 20 point scale of the test. Higher scores indicate worse delirium.
Time Frame: Baseline, day of surgery (twice), post-operative days 1 - 5 (twice), 6 weeks +/- 3 weeks
Population: Subjects who completed surgery on protocol and had at least 1 postoperative CAM-3D assessment performed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | CN-105 | Placebo
Number analyzed (Participants) | 135 | 48
score on a scale | 1 [1 to 2] | 2 [1 to 2]
Statistical Analysis 1: Comparison: CN-105 vs Placebo; Test type: Other; p = 0.189, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Surgery to 6-week follow-up visit
Description: Hospital records were reviewed for any CTCAE (v5.0) events rated grade II or higher during index hospitalization or reported to study team members during study follow-up visits.
Arm/Group | CN-105 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/49
Serious Adverse Events (participants affected / at risk) | 11/137 | 11/49
Other Adverse Events (participants affected / at risk) | 105/137 | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CN-105 (N=137) | Placebo (N=49)
ANEMIA (Blood and lymphatic system disorders) | 1 | 3
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
CYSTOSCOPY FOR REMOVAL OF URINARY CATHETER (Surgical and medical procedures) | 0 | 1
DELIRIUM (Psychiatric disorders) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0
FATIGUE (General disorders) | 0 | 1
GASTRIC STENOSIS (Gastrointestinal disorders) | 0 | 1
HEART FAILURE EXACERBATION (Cardiac disorders) | 1 | 0
HEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 3
HYPOXEMIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
ILEUS (Gastrointestinal disorders) | 1 | 0
INTRAOPERATIVE ARTERIAL INJURY (Injury, poisoning and procedural complications) | 1 | 0
LARYNGEAL EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
MEDICAL PROCEDURE (Surgical and medical procedures) | 2 | 1
MOBITZ TYPE 1 AV BLOCK (Cardiac disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0
NEOPLASM (METASTATIC SQUAMOUS CELL LUNG CANCER) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PHARYNGITIS/OTALGIA (Infections and infestations) | 0 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
POST-OPERATIVE ILEUS (Gastrointestinal disorders) | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CN-105 (N=137) | Placebo (N=49)
ABDOMINAL MASS (Injury, poisoning and procedural complications) | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 4 | 1
ALT INCREASED (Investigations) | 1 | 0
ANEMIA (Blood and lymphatic system disorders) | 30 | 9
ANOREXIA (Metabolism and nutrition disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
AST INCREASED (Investigations) | 3 | 0
BLADDER SPASM (Renal and urinary disorders) | 0 | 1
CEREBROSPINAL FLUID LEAKAGE. (Nervous system disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 3 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 1
CREATININE INCREASE (Investigations) | 5 | 0
CYSTITIS NONINFECTIVE (VS PROSTATITIS, DYSURIA, PROTEINURIA) (Renal and urinary disorders) | 1 | 0
DECREASED LYMPHOCYTE COUNT (Investigations) | 27 | 15
DECREASED PLATELET COUNT (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 2 | 2
DEPRESSION (IE ADJUSTMENT DISORDER WITH ANXIETY AND DEPRESSED MOOD) (Psychiatric disorders) | 0 | 1
DIARRHEA (Gastrointestinal disorders) | 3 | 2
DIZZINESS (Nervous system disorders) | 3 | 5
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EGD (Surgical and medical procedures) | 1 | 0
EPIDIDYMO-ORCHITIS (Infections and infestations) | 0 | 1
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 | 0
ERYTHEMATOUS AREA NOTED IN THE RIGHT ANTECUBITAL FOSSA (Skin and subcutaneous tissue disorders) | 0 | 1
ESOPHAGEAL ULCER (Gastrointestinal disorders) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
FASCIAL DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
FATIGUE (General disorders) | 3 | 0
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 | 1
FEVER (General disorders) | 2 | 0
FLU LIKE SYMPTOMS (General disorders) | 1 | 0
GASTROESOPHAGEAL REFLUX- (Gastrointestinal disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 1
HEMATURIA (Renal and urinary disorders) | 1 | 1
HEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HIGH CHEST TUBE OUTPUT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPERBILIRUBINEMIA (Investigations) | 0 | 1
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 | 6
HYPERKALEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPERTENSION (Vascular disorders) | 61 | 22
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 11 | 4
HYPOCALCEMIA (Metabolism and nutrition disorders) | 10 | 3
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 2 | 1
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOTENSION (Vascular disorders) | 12 | 3
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 5 | 2
ILEUS (Gastrointestinal disorders) | 1 | 1
INCREASED CREATININE (Investigations) | 0 | 1
INFECTION (Infections and infestations) | 17 | 6
INFUSION SITE EXTRAVASATION (General disorders) | 2 | 0
INR INCREASED (Investigations) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 1
IV INFILTRATION (General disorders) | 0 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 2 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0
LOW ALBUMIN (Metabolism and nutrition disorders) | 1 | 1
LOW LYMPH COUNT (Investigations) | 1 | 0
LOW URINE OUTPUT (Investigations) | 1 | 0
MALAISE (General disorders) | 1 | 0
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 | 0
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 1
NAUSEA (Gastrointestinal disorders) | 6 | 4
NON-INFECTIVE CYSTITIS (Renal and urinary disorders) | 1 | 0
OPERATIVE REPAIR OF EVISCERATION OF BOWEL FROM MIDLINE INCISION (Surgical and medical procedures) | 1 | 0
PAIN (Gastrointestinal disorders) | 1 | 2
PAIN (General disorders) | 7 | 3
PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
PAIN (Reproductive system and breast disorders) | 1 | 0
PAROTITIS (Infections and infestations) | 0 | 1
PERMANENT PACEMAKER PLACEMENT (Surgical and medical procedures) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
POSSIBLE HYPOTHYROIDISM (Endocrine disorders) | 1 | 0
POST-OPERATIVE ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
PRURITIS (Skin and subcutaneous tissue disorders) | 2 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RADICULITIS (Nervous system disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RIGHT INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
SEVERE PROTEIN CALORIE MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
SHOULDER INJECTION (Surgical and medical procedures) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 2 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 3 | 0
SYNCOPE (Nervous system disorders) | 1 | 2
TRANSFER TO LONG-TERM CARE FACILITY DUE TO MENTAL ACUITY CONCERN (Social circumstances) | 1 | 0
UNPLANNED SURGICAL PROCEDURE (Surgical and medical procedures) | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 3
URINARY RETENTION (Renal and urinary disorders) | 4 | 3
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 2 | 0
URINARY URGENCY (Renal and urinary disorders) | 0 | 1
URINE OUTPUT DECREASED (Investigations) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
VASOVAGAL REACTION (Nervous system disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 5 | 5
VULVOVAGINAL ATROPHY/VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03802396/Prot_SAP_000.pdf